CLINICAL TRIAL: NCT04189874
Title: Efficacy of BioFire FilmArray Gastrointestinal Panel (FGP) to Reduce Hospital Costs Associated With Contact Isolation
Brief Title: Stool Testing With Molecular Assay to Minimize Contact Precautions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Giulio DiDiodato (Other)
Collaborators: Biomerieux inc (Industry)
Responsible Party: Sponsor-Investigator, Giulio DiDiodato, Chief Research Scientist, Royal Victoria Hospital, Canada
Organization: Royal Victoria Hospital, Canada (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: REB#R19-031
Record Dates: First submitted 2019-12-01; First posted 2019-12-06 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Infectious Gastroenteritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional stool testing (Active Comparator): All patients randomly allocated to this arm will have their stools tested for the following:
  a) Bacterial culture for Salmonella, Shigella, E.coli O157 and Campylobacter - specimen in Enteric Pathogen Transport medium (EPT) planted to: i) MacConkey agar, Sorbitol-MacConkey agar, Hektoen agar and Selenite broth all incubated overnight at 350C ii) Campylobacter agar incubated for 48 hours at 420C in a microaerophilic atmosphere b) Bacterial culture for Yersinia (≤ 18 years old): EPT specimen sent to Dynacare Laboratories for processing, results back in 10-14 days c) Ova & Parasites investigation: Sodium acetate-Acetic Acid-Formalin specimen sent to the Public Health Laboratories (PHL) for testing, results back in 7-10 days d) Viral culture: rarely requested, requires a specimen in a sterile container, sent to the PHL for testing, results back in 5-7 days e) Clostridioides difficile: specimen in sterile container, results in 1h (GeneXpert)
  Interventions: Diagnostic Test: Conventional Stool Testing
- BioFire FilmArray Gastrointestinal Panel (Experimental): All patients randomly allocated to this arm will have their stools tested using a PCR-based molecular assay that can simultaneously test for 22 different infectious pathogens with a turnaround time of approximately 1 hour. As results become available, they will be available for review by the patient's healthcare providers in the electronic medical record.
  Interventions: Diagnostic Test: BioFire FilmArray Gastrointestinal Panel

INTERVENTIONS:
Diagnostic Test: Conventional Stool Testing — Stools are tested using conventional culture techniques
  Arms: Conventional stool testing
Diagnostic Test: BioFire FilmArray Gastrointestinal Panel — Molecular-based stool assay
  Arms: BioFire FilmArray Gastrointestinal Panel

SUMMARY:
This study evaluates the impact of infectious diseases molecular-based stool testing compared to conventional stool testing on reducing the need for contact precautions among hospitalized patients. Half of patients' stools will be tested with the molecular assay , while the other half will be tested with conventional testing.

DETAILED DESCRIPTION:
Acute infectious gastroenteritis can be caused by viruses, bacteria or parasites, resulting in a diarrheal illness that may be accompanied by fever, abdominal pain and/or cramping, hematochezia, nausea, and vomiting. Up to 12.5% to 25% of the population develop a gastrointestinal infection each year, with the majority of cases being self-limiting and symptoms usually resolving within 14 days without treatment. While the vast majority of the estimated 4 million Canadians who develop gastroenteritis have a mild and self-limited illness, approximately 9 250 to 14 150 are hospitalized each year with 1.6% to 2.2% dying from their disease.

For hospitalized patients, the majority will have stool samples collected and tested using standard microbiology methods that includes culture for bacteria, nucleic acid amplification for viruses and bacteria and microscopy or enzyme immunoassays for parasites. The number of pathogens that can be identified is limited in most microbiology laboratories, and the turnaround time to reporting can take up to 3 days. Recently, new nucleic acid amplification technologies have been developed that can test for multiple gastrointestinal pathogens in a single run that usually takes less than a 1 day turnaround time to reporting.

The BioFire® FilmArray Gastrointestinal Panel (FGP) is a multiplex polymerase chain reaction test that can simultaneously test for 22 different viruses, bacteria and parasites with excellent sensitivity and specificity with a turnaround time of 1 hour. Compared to conventional testing methods, the FGP costs 40% more, or about $180 (CDN) per test. Despite detecting more pathogens in a shorter period of time, a recent systematic review did not find any evidence to support a positive impact on either improved patient outcomes or cost-effectiveness compared to conventional testing. Since most gastrointestinal illness episodes are mild and self-limiting, it may not be feasible to design a randomised trial to demonstrate clinical efficacy of test-treatment given the majority of the 22 pathogens detected by the FGP do not benefit from antimicrobial therapy. Instead, measuring other outcomes like reduced utilization of hospital resources such as contact isolation days, could provide evidence for both clinical benefit and cost-effectiveness.

To date, the available evidence on the cost-effectiveness of the FGP assay has been based largely on observational studies, usually historically controlled before-after designs associated with high risk of bias. The only study that was of sufficient quality to be included in a systematic review of cost-effectiveness utilized a different PCR-based test. Since the FGP assay has been shown to have very similar diagnostic characteristics in a head-to-head comparison with this other PCR-based assay, the results will be used to inform the primary outcome for this study. In the study by Goldenberg et al., differences in contact isolation days between conventional (observed) and PCR-based testing (simulated) were estimated and found to result in a reduction of 34.3% in contact isolation days in the PCR-based group. Among the 800 patients, this amounted to a mean reduction of 0.94 contact isolation days per patient. Unfortunately, confidence intervals were not estimated for this point estimate. The cost of a single isolation day was reported as approximately £88 (UK) for fiscal 2011/2012. A breakeven analysis demonstrated that a reduction of 252 contact isolation days, a reduction of 11.4%, was needed to offset the increased costs associated with the PCR-based assay. The cost of the PCR-based assay used in this study was 0.4 times the cost of the FGP assay, suggesting that the number of contact isolation days needed to breakeven with the FGP assay could be as high as 635. In a more recent conference report of a randomised study in the United Kingdom using FGP, an interim analysis estimated a reduction in contact isolation days by 0.9 days per patient (95% CI 0.4 to 1.6). There was no data provided for cost-effectiveness. Given the extent of uncertainty around both the clinical effectiveness and cost-effectiveness of the FGP assay, a randomised test-treat trial would be the best option to resolve these uncertainties.

ELIGIBILITY:
Inclusion Criteria:

* Any patient in whom an appropriate stool sample has been collected and received by the microbiology laboratory that is:

  1. accompanied by a physician request for microbiologic testing for viruses, bacteria and/or parasites, and is
  2. appropriate for testing as determined by the microbiology laboratory standard (stool sample must have sufficient consistency to take shape of collection container), and
  3. patient is admitted to hospital
  4. Stool testing done between Monday 08:00 and Friday 14:00 a. The Infection Prevention and Control Practitioners (IPAC) are only available to review the stool test results between Monday 08:00 and Friday 17:00. Since IPAC is responsible for all decisions regarding contact isolation initiation and discontinuation, time delays from stool test reporting and decisions regarding contact isolation on the weekends or after 17:00 on weekdays would confound the primary outcome. As a result, FGP testing will only be available between Monday 08:00 and Friday 14:00 during the study period since each FGP test requires approximately 1 hour to complete, and the laboratory can only run 1 test at a time. Outside these hours, only conventional testing will be available.

Exclusion Criteria:

1. Immunocompromised patients
2. Investigation of possible diarrheal outbreak by either public health officials or infection prevention and control practitioners
3. Nosocomial Clostridioides difficile infection defined as a positive polymerase chain reaction test in any patient who meets any of the following criteria:

   1. Has been hospitalized for ≥ 72 hours and then develops ≥ 3 loose bowel movements per day
   2. Develops ≥ 3 loose bowel movements per day regardless of length of hospital stay and has been hospitalized in the preceding 3 months for ≥ 48 hours

Ages: 1 Month to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2019-12-18 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-02-12 (Actual)

PRIMARY OUTCOMES:
Mean difference in hospital costs associated with contact isolation | up to 1 year
  Direct hospital costs associated with contact isolation such as personal protective equipment, terminal cleaning, etc.. will be estimated for each arm and their mean difference estimated

SECONDARY OUTCOMES:
1. Mean difference in costs associated with differences in antimicrobial utilization | up to 1 year
  Mean difference in costs between arms associated with antimicrobial utilization
2. Difference in proportion of patients with any change in empiric antimicrobial treatment | up to 1 year
  differences in proportion of patients with any change in antibiotic therapy as a result of molecular assay
3. Mean difference in costs associated with differences in diagnostic imaging utilization | up to 1 year
  Mean difference in costs associated with diagnostic imaging between arms
4. Mean differences in costs associated with differences in endoscopy utilization | up to 1 year
  Mean differences in costs associated with endoscopic utilization between arms
5. Mean difference in total costs associated with the composite outcome of (hospital days + antimicrobials + diagnostic imaging + endoscopy + contact isolation) | up to 1 year
  Mean differences in total costs associated with overall utilization differences between arms
6. Ranking of responses to 2-item questionnaire assessing physician perceptions of value of PCR-based assay using a 5-point Likert scale. | up to 1 year
  Each physician will be asked to rank how much they agree/disagree with the following statements using a Likert scale (1=strongly disagree, 2=moderately disagree, 3=neither disagree nor agree, 4=moderately agree, 5=strongly agree)
  1. Without the earlier results provided by the FGP assay, my patient would have experienced possible/probable harm
  2. Because of the earlier results provided by the FGP assay, my patient's treatment plan was changed (for example, change or discontinuation of antibiotic treatment, discontinuation of contact isolation, earlier discharge from hospital)

CONTACTS AND LOCATIONS:
Overall Officials: Giulio DiDiodato, PhD, Principal Investigator — Royal Victoria Regional Health Centre
Locations (1):
- Royal Victoria Regional Health Centre, Barrie, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Excel csv of anonymized IPD - all data collected will be shared
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data will become available after study recruitment closed and data has been cleaned. Data will be available indefinitely afterwards.
Access Criteria: Email request